CLINICAL TRIAL: NCT01587534
Title: Phase 2 Study of Randomized Controlled Trial of Pancreatic Enzyme Supplementation in Patients With Unresectable Pancreatic Cancer
Brief Title: Pancreatic Enzyme Supplementation in Patients With Unresectable Pancreatic Cancer (PESUP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Pharmbio Korea Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Sang Myung Woo, Staff physician, Ceneter for Liver Cancer, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCCCTS-11-570
Record Dates: First submitted 2012-04-25; First posted 2012-04-30 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Pancreatic Cancer
Keywords: Unresectable Pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- pancreatic enzyme replacement therapy (Experimental): The pancreatic enzyme preparation under investigation is Norzyme ® 6 - 9 tablets per day.
  Interventions: Drug: Norzyme
- Placebo (No Intervention): The placebo will match the active drug in appearance, taste, and weight and contained pharmacologically inactive substances.

INTERVENTIONS:
Drug: Norzyme — Patients will be randomized to receive either pancreatic enzyme replacement therapy or placebo. Patients will use two capsules three times daily during main meals and one capsule three times daily during in between snacks. The pancreatic enzyme preparation under investigation is Norzyme ® 6 - 9 tablets per day.
  Other Names: placebo
  Arms: pancreatic enzyme replacement therapy

SUMMARY:
The investigators planned a prospective, randomized, placebo controlled trial to test the hypothesis that weight loss in patients with unresectable pancreatic cancer with occlusion of the pancreatic duct can be reduced or prevented by pancreatic enzyme replacement therapy in combination with dietary counseling.

DETAILED DESCRIPTION:
Pancreatic cancer has the worst overall prognosis with fewer than 3% of affected patients alive ﬁve years after the initial diagnosis. It is the fourth leading cause of death from cancer in Korea. 80-90% of patients have locally unresectable or advanced metastatic disease and for these patients only palliative treatment options remain. Symptoms include obstructive jaundice, duodenal obstruction, pain, and weight loss. Palliative treatment is mainly directed against the former three. Interventions to prevent (further) weight loss have as yet received little or no attention, in spite of the frequent occurrence of this symptom. About 90% of patients with pancreatic carcinoma have weight loss at the time of diagnosis. In addition, Weight loss prior to chemotherapy was found to have a prognostic effect on survival in a range of different tumor types.

There is a limited range of studies investigating the incidence of exocrine insufficiency in pancreatic cancer. Studies available indicate a high incidence of exocrine insufficiency in unresectable pancreatic cancer patients and patients before and after pancreatic cancer surgery. The previous reports showed that 68-92% of pancreatic cancer patients were exocrine insufficient. Such high incidences of exocrine insufficiency in pancreatic cancer patients support the use of pancreatic enzyme replacement therapy in this patient group. The guidelines for the management of patients with pancreatic cancer periampullary and ampullary carcinoma published in Gut promote the use of pancreatic enzyme replacement therapy to maintain weight and to increase quality of life in this patient group. However, studies evaluating the efficacy of pancreatic enzyme replacement therapy in pancreatic cancer are lacking to date. There have been no systematic reviews and only one randomized control trial involving a small sample of 21 patients with unresectable cancer of the pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for inclusion, each patient must fulfill each of the following criteria:

  1. Subjects with unresectable pancreatic cancer preferably proven by cytology or histology
  2. not eligible for surgery because of poor general condition, local unresectability, or advanced disease with metastases
  3. Age over 18 years old
  4. Performance status (ECOG scale): 0-2
  5. Agree to record daily food intake
  6. Patients should sign a written informed consent before study entry

Exclusion Criteria:

* Patients will be excluded from the study for any of the following reasons:

  1. History of major gastrointestinal surgery
  2. history of chronic gastrointestinal disease (for example, Crohn's disease)
  3. Diabetes decompensated
  4. Diabetes mellitus with severe gastroparesis
  5. presence of pancreatic pseudocysts impeding gastric or duodenal passage
  6. any use of antacids, mucosal protective agents, H 2 receptor antagonists, or proton pump inhibitors that could not be discontinued
  7. concomitant medication affecting gastroduodenal motility (e.g. metoclopramide and erythromycin), or interfering with bile secretion (e.g. bile acids)
  8. Abusive use of alcohol in the three months preceding the study;
  9. known allergy to pancreatin
  10. Any major surgery within 4 weeks prior to study treatment
  11. Pregnant or lactating woman
  12. Any patients judged by the investigator to be unfit to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
the change in body weight at eight weeks after the randomisation | at baseline and 4, 8 week, 24 week
  the percentage change in body weight at eight weeks after the randomisation

SECONDARY OUTCOMES:
Frequency and intensity of abdominal pain daily | at baseline and 4, 8 week, 24 week
Frequency of bowel movements per day | at baseline and 4, 8 week, 24 week

CONTACTS AND LOCATIONS:
Overall Officials: Sangmyung Woo, M.D, Principal Investigator — National Cancer Center
Locations (1):
- NATIONAL CANCER CENTER 323, Ilsan-ro, Ilsandong-gu,, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Woo SM, Joo J, Kim SY, Park SJ, Han SS, Kim TH, Koh YH, Chung SH, Kim YH, Moon H, Hong EK, Lee WJ. Efficacy of pancreatic exocrine replacement therapy for patients with unresectable pancreatic cancer in a randomized trial. Pancreatology. 2016 Nov-Dec;16(6):1099-1105. doi: 10.1016/j.pan.2016.09.001. Epub 2016 Sep 4. PMID 27618657